CLINICAL TRIAL: NCT02850328
Title: Muscular Force Generation in Microgravity (ForceGeneration)
Brief Title: Muscular Force Generation in Microgravity
Acronym: ForceGeneratio
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Collaborators: Novespace (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2014-A00814-43
Record Dates: First submitted 2016-04-21; First posted 2016-08-01 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2016-07

CONDITIONS: Maximum Voluntary Contraction
MeSH Terms: interventions — Weightlessness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- high-load resistance training for long term space flights (Other): Short duration electrical will be delivered and the resulting EMG will be recorded. Intensity of electrical stimulation will be progressively increased until we observed a maximal EMG response.
  Finally an ultrasound probe (similar to that used for prenatal diagnostic imaging) will be fixed behind your calf in order to visualize muscle.
  Interventions: Other: examination of muscle function and MVC in weightlessness

INTERVENTIONS:
Other: examination of muscle function and MVC in weightlessness — MVC tested during three different tasks: (1) leg press, (2) plantarflexion and (3) grip strength.
  parameters of muscle function that can be easily implemented in parabolic flight:
  * Rate of force development
  * Electromyographic activity
  * Ultrasound measure: fascicle length and pennation angle of the gastrocnemius medialis muscle
  * Superimposed twitch torque (M-waves at rest and V-waves in MVC conditions)
  * Maximum voluntary activation capacity (%VA): %VA = (1-[torque superimposed twitch/torque resting twitch])*100%.

SUMMARY:
The aim of this study is to evaluate the applicability of high-load resistance training as a countermeasure for long term space flights, the current project has two scientific goals.

The main objective is to perform a deeper examination of muscle function and MVC in weightlessness (parabolic flight).

The secondary objective is to gather further insight into the underlying mechanisms and structures based on investigations targeting the neuromuscular and musculotendinous systems and their interaction.

DETAILED DESCRIPTION:
The findings from water immersion indicated that some motor tasks, such as plantarflexion (25), but not others, such as the leg-press (7), appear to be affected. Thus, it would be relevant to test a number of motor tasks and body regions. On the other hand, parabolic flight requires that methodologies can be performed in a quick efficient fashion. Hence, we propose examining ankle plantarflexion, leg-press and grip-force.

The primary hypothesis is that plantarflexion MVC will be reduced in the microgravity phase of parabolic flight.

As secondary parameters will be assessed parameters of muscle function that can be easily implemented in parabolic flight, such as electromyography and ultrasound measurements of the musculotendinous unit. To assess the muscular system more deeply, for plantarflexion superimposed twitches will be performed (16) during MVC and at rest. An additional experimental condition placing foam (unstable surface; standard size) under the foot during plantarflexion will be included. This approach increases the challenge for the neuromuscular control system and, under such conditions, MVC is reduced (29).

These secondary investigations, which do not prohibitively complicate the practical implementation of the project, will help to understand what is happening in the musculature should we indeed find impediments of muscle force generation in microgravity.

The aim of this study is to evaluate the applicability of high-load resistance training as a countermeasure for long term space flights, the current project has two scientific goals.

The main objective is to perform a deeper examination of muscle function and MVC in weightlessness (parabolic flight).

The secondary objective is to gather further insight into the underlying mechanisms and structures based on investigations targeting the neuromuscular and musculotendinous systems and their interaction.

The main judgment criteria is the MVC tested during three different tasks: (1) leg press, (2) plantarflexion and (3) grip strength.

As secondary criteria, we will assess parameters of muscle function that can be easily implemented in parabolic flight:

* Rate of force development
* Electromyographic activity
* Ultrasound measure: fascicle length and pennation angle of the gastrocnemius medialis muscle
* Superimposed twitch torque (M-waves at rest and V-waves in MVC conditions)
* Maximum voluntary activation capacity (%VA): %VA = (1-[torque superimposed twitch/torque resting twitch])*100%.

The primary hypothesis is that plantarflexion and knee extension force generation capacity will be reduced, but not grip-force, in the microgravity phase of parabolic flight.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (men or women)
* Aged from 21 to 65
* Affiliated to a Social Security system and, for non-French resident, holding a European Health Insurance Card (EHIC)
* Who accepted to take part in the study
* Who have given their written stated consent
* Who have their right leg as their preferred leg
* Who has passed a medical examination similar to a standard aviation medical examination for private pilot aptitude (JAR FCL3 Class 2 medical examination). There will be no additional test performed for subject selection.

Subjects will be staff member of the team or of other teams participating in the parabolic flight campaign

Exclusion Criteria:

* Person who took part in a previous biomedical research protocol, of which exclusion period is not terminated
* Person with orthopaedic disorders in the upper or lower limbs
* Person with neurological disorders
* Pregnant women

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2014-09; Primary Completion 2017-09 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
maximum voluntary contraction (MVC) | baseline
  tested during three different tasks: (1) leg press, (2) plantarflexion and (3) grip strength.

SECONDARY OUTCOMES:
parameters of muscle function, Rate of force development | baseline
parameters of muscle function, Electromyographic activity | baseline
parameters of muscle function, Ultrasound measure: fascicle length | baseline
parameters of muscle function, Ultrasound measure: pennation angle of the gastrocnemius medialis muscle | baseline
parameters of muscle function, Superimposed twitch torque (M-waves at rest and V-waves in MVC conditions) | baseline
parameters of muscle function, Maximum voluntary activation capacity (%VA): %VA = (1-[torque superimposed twitch/torque resting twitch])*100%. | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Pierre DP Denise, PhD, Principal Investigator — UMR 1075 UFR de Médecine Caen
Locations (1):
- Caen CHU, Caen, France

IPD SHARING:
Plan to Share IPD: No